CLINICAL TRIAL: NCT04340115
Title: Special Drug Use - Results Survey Of Evaluating Safety And Effectiveness Of RINVOQ In Patients With Rheumatoid Arthritis
Brief Title: Study To Assess Frequency Of Serious Infections In Clinical Practice In Japan For Adult Participants With Rheumatoid Arthritis Receiving Oral RINVOQ Tablets
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P19-565
Record Dates: First submitted 2020-04-07; First posted 2020-04-09 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Rheumatoid Arthritis (RA); RINVOQ; Upadacitinib; ABT-494
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants treated with RINVOQ: Participants treated with upadacitinib in accordance with approved local label. Decision to treat with upadacitinib was made prior to offering participation in this study.

SUMMARY:
Rheumatoid Arthritis (RA) is a chronic inflammatory disease causing pain, stiffness, swelling and loss of joint function. RA can reduce the ability to perform everyday tasks. The purpose of this study is to observe the incidence of serious infections, regardless of their relationship to RINVOQ, in Japanese daily practice.

RINVOQ is an approved drug for the treatment of adults with moderately to severely active RA. This study evaluates medical records from institutions participating in the study to identify any adverse events (untoward medical occurrence), and reasons for discontinuation of RINVOQ in participants taking the study drug. A target of 1000 Japanese participants' data will be observed for 3 years.

Participants will receive RINVOQ per their physicians' usual prescription. Individual data will be collected for three years.

No additional study-related tests will be conducted during routine clinic visits. Only data which are routinely collected during clinic visits will be utilized for this study.

ELIGIBILITY:
Inclusion Criteria:

- All participants treated with RINVOQ.

Exclusion Criteria:

- Participants not taking RINVOQ.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult participants with rheumatoid arthritis according to local label.
Sampling Method: Non-Probability Sample
Enrollment: 4211 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Number (Percentage) Of Participants Who Reported Of Serious Infection | 24 Weeks
  Number (Percentage) of participants with incidence of serious infections are reported.

SECONDARY OUTCOMES:
Number (Percentage) Of Participants Who Reported Adverse Drug Reactions (ADRs) | 24 Weeks
  Number (Percentage) of participants who report ADRs. An untoward medical occurrence in a participant, called an adverse event (AE) whose causal relationship with the product cannot be ruled out is considered an ADR.
Number (Percentage) Of Participants Who Reported Of Serious Infection | 3 Years
  Number (Percentage) of participants with incidence of serious infections are reported.
Number (Percentage) Of Participants Who Reported Malignancies | 3 Years
  Number (Percentage) of participants with incidence of malignancies are reported.
Number (Percentage) Of Participants Who Reported Major Adverse Cardiovascular Events (MACE) | 3 Years
  Number (Percentage) of participants with incidences of MACE are reported.
Number (Percentage) Of Participants Who Reported Venous Thrombosis And Pulmonary Embolus (VTEs) | 3 Years
  Number (Percentage) of participants with incidences of VTEs are reported.
Percentage Of Participants Achieving Clinical Remission (CR) on Disease Activity Score-28 With C-Reactive Protein (DAS28-CRP) | 24 Weeks
  CR is defined as DAS28 CRP <2.6. The Disease Activity Score (DAS) 28 is a validated index of rheumatoid arthritis disease activity. Scores on the DAS28 range from 0 (lowest disease activity) to 10 (highest disease activity).
Percentage Of Participants Achieving Low Disease Activity (LDA) on Disease Activity Score-28 With C-Reactive Protein (DAS28-CRP) | 24 Weeks
  LDA is defined as DAS 28-CRP >= 2.6 but < 3.2. The Disease Activity Score (DAS) 28 is a validated index of rheumatoid arthritis disease activity. Scores on the DAS28 range from 0 (lowest disease activity) to 10 (highest disease activity).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1017):
- Japan (1017):
  - Kanda Orthopedics & Rheumatology Clinic /ID# 238592, Gamagōri, Aichi-ken
  - Handa City Hospital /ID# 232198, Handa-shi, Aichi-ken
  - Handa City Hospital /ID# 244106, Handa-shi, Aichi-ken
  - Ichinomiya Orthopedic /ID# 226814, Ichinomiya-shi, Aichi-ken
  - Ichinomiya Municipal Hospital /ID# 251000, Ichinomiya-shi, Aichi-ken
  - Haimoto Clinic /ID# 243718, Kasugai, Aichi-ken
  - Kasugai Orthopaedic Clinic /ID# 239041, Kasugai-shi, Aichi-ken
  - Sanjinkai Asahi Hospital /ID# 242397, Kasugai-shi, Aichi-ken
  - Kurotsuchi Orthopaedic Clinic /ID# 224194, Kasugashi, Aichi-ken
  - Kurotsuchi Orthopaedic Clinic /ID# 233900, Kasugashi, Aichi-ken
  - Komaki Chiba Orthopedics Clinic /ID# 233960, Komaki-shi, Aichi-ken
  - Komaki City Hospital /ID# 232586, Komaki-shi, Aichi-ken
  - Komaki Yotei Memorial Hospital /ID# 229104, Komaki-shi, Aichi-ken
  - Ueda Orthopedic Surgical Clinic /ID# 232359, Konan-chi, Aichi-ken
  - Asano Orthopedic Clinic /ID# 224110, Konan-shi, Aichi-ken
  - Sankuro Hospital /ID# 233952, Kozakacho, Aichi-ken
  - Aichi Medical University Hospital /ID# 224009, Nagakute, Aichi-ken
  - Aichi Medical University Hospital /ID# 224995, Nagakute, Aichi-ken
  - Japanese Red Cross Aichi Medical Center Nagoya Daiichi Hospital /ID# 279485, Nagoya, Aichi-ken
  - Arako Clinic /ID# 229654, Nagoya, Aichi-ken
  - Nagoya Kyoritsu Hospital /ID# 231712, Nagoya, Aichi-ken
  - Sato Orthopedic Clinic /ID# 231726, Nagoya, Aichi-ken
  - Japan Organization of Occupational Health and Safety Chubu Rosai Hospital /ID# 225310, Nagoya, Aichi-ken
  - Juko Memorial Hospital /ID# 238602, Nagoya, Aichi-ken
  - Daido Clinic - Nagoya /ID# 239032, Nagoya, Aichi-ken
  - Minami Medical Health Cooperative /ID# 275121, Nagoya, Aichi-ken
  - NHO Nagoya Medical Center /ID# 229655, Nagoya, Aichi-ken
  - Hashimoto Orthopedic Clinic /ID# 225347, Nagoya, Aichi-ken
  - Moriyama Itsuki Hospital /ID# 231745, Nagoya, Aichi-ken
  - Nagoya City University East Medical Center /ID# 238530, Nagoya, Aichi-ken
  - Nagoya City University East Medical Center /ID# 239399, Nagoya, Aichi-ken
  - Saito Clinic /ID# 223262, Nagoya, Aichi-ken
  - Kawana Hospital /ID# 222583, Nagoya, Aichi-ken
  - Sugiura Internal Medicine Clinic /ID# 227627, Nagoya, Aichi-ken
  - Nagoya University Hospital /ID# 231716, Nagoya, Aichi-ken
  - Nagoya City University Hospital /ID# 232357, Nagoya, Aichi-ken
  - National Center for Geriatrics and Gerontology /ID# 240937, Obu-shi, Aichi-ken
  - Uno Orthopedic Clinic /ID# 227640, Okazaki-shi, Aichi-ken
  - Aichi Medical University Medical Center /ID# 255162, Okazaki-shi, Aichi-ken
  - Kato Orthopedic Clinic /ID# 223263, Okazaki-shi, Aichi-ken
  - Arakawa Medical Clinic /ID# 224994, Owariashi-shi, Aichi-ken
  - Jyunshinkai Inoue Hospital /ID# 233853, Seto-shi, Aichi-ken
  - Nishichita General Hospital /ID# 252178, Tokai-shi, Aichi-ken
  - Fujita Health University Hospital /ID# 226743, Toyoake, Aichi-ken
  - National Hospital Organization Toyohashi Medical Center /ID# 239042, Toyohashi, Aichi-ken
  - National Hospital Organization Toyohashi Medical Center /ID# 244697, Toyohashi, Aichi-ken
  - Fukui Clinic /ID# 223311, Toyohashi, Aichi-ken
  - Aoyama Hospital /ID# 233897, Toyokawa, Aichi-ken
  - Kasai Orthopedic Surgical Clinic /ID# 233899, Toyokawa, Aichi-ken
  - Sasaki Orthopedic Surgical Clinic /ID# 233951, Toyokawa, Aichi-ken
  - Toyota Memorial Hospital /ID# 232197, Toyota-shi, Aichi-ken
  - Funahashinaika Clinic /ID# 222605, Toyota-shi, Aichi-ken
  - Kainan Hospital /ID# 251696, Yatomi-shi, Aichi-ken
  - Hikosaka Surgery Clinic /ID# 241064, 津島市, Aichi-ken
  - Akita Renal, Collagen and Rheumatology disease Clinic /ID# 238580, Akita, Akita
  - Akita City Hospital /ID# 258322, Akita, Akita
  - Akita University Hospital /ID# 262657, Akita, Akita
  - Nakadori General Hospital /ID# 249517, Akita, Akita
  - Odate Municipal General Hospital /ID# 225774, Odate-shi, Akita
  - Akita Rosai Hospital /ID# 243722, Odate-shi, Akita
  - Hiraka General Hospital /ID# 269114, Yokote, Akita
  - Hiraka General Hospital /ID# 261252, Yokote-shi, Akita
  - JA Akita Koseiren Yuri Union General Hospital /ID# 238595, Yurihonjo-shi, Akita
  - Aomori Prefectural Central Hospital /ID# 226735, Aomori, Aomori
  - Aomori Jikeikai Hospital /ID# 268346, Aomori, Aomori
  - Tsugaru General Hospital /ID# 222610, Goshogawara-shi, Aomori
  - Kanagi Hospital /ID# 265630, Goshogawara-shi, Aomori
  - Nakazawa Sports Clinic /ID# 230217, Hachinohe-shi, Aomori
  - Aomori Rosai Hospital /ID# 229158, Hachinohe-shi, Aomori
  - Hirosaki Station Clinic /ID# 266722, Hirosaki-shi, Aomori
  - Kaneko Orthopedic Surgical Clinic /ID# 224955, Hirosaki-shi, Aomori
  - Hirosaki University Hospital /ID# 238581, Hirosaki-shi, Aomori
  - Mutsu General Hospital /ID# 267370, Mutsu, Aomori
  - Satoru Orthopedic Clinic /ID# 225866, Towada-shi, Aomori
  - Asahi General Hospital /ID# 226832, Asahi, Chiba
  - Tsuchida Clinic /ID# 225309, Chiba, Chiba
  - Chiba Aoba Municipal Hospital /ID# 229039, Chiba, Chiba
  - Chiba University Hospital /ID# 230289, Chiba, Chiba
  - Chiba University Hospital /ID# 238878, Chiba, Chiba
  - Yonemoto Orthopedic Surgical Clinic /ID# 224600, Chosei-gun, Chiba
  - Chiba Rosai Hospital /ID# 232580, Ichihara-shi, Chiba
  - Yarita Hospital /ID# 256196, Ichihara-shi, Chiba
  - Shirogane Orthopedic Surgery Hospital /ID# 229037, Ichihara-shi, Chiba
  - Hidaka Clinic /ID# 240660, Ichihara-shi, Chiba
  - Teikyo University Chiba Medical Center /ID# 238472, Ichihara-shi, Chiba
  - Ito Clinic /ID# 248812, Ichikawa-shi, Chiba
  - Tokyo Dental College Ichikawa General Hospital /ID# 256181, Ichikawa-shi, Chiba
  - Kamagaya General Hospital /ID# 247769, Kamagaya-shi, Chiba
  - Kameda General Hospital /ID# 233873, Kamogawa-shi, Chiba
  - The Jikei University Kashiwa Hospital /ID# 269113, Kashiwa, Chiba
  - Kashiwa Hasegawa Orthopaedics /ID# 244208, Kashiwa, Chiba
  - Tomita Clinic /ID# 223310, Kashiwa-shi, Chiba
  - Asunaro Clinic /ID# 243687, Kimitsu, Chiba
  - Gengendo Kimitsu Hospital /ID# 244098, Kimitsu-shi, Chiba
  - Kisarazu Toho Hospital /ID# 224474, Kisarazu-shi, Chiba
  - Kisarazu Toho Hospital /ID# 238543, Kisarazu-shi, Chiba
  - Kazusa Orthopedic Surgical Clinic /ID# 260730, Kisarazu-shi, Chiba
  - MiruMiru Clinic /ID# 258328, Kisarazu-shi, Chiba
  - Kimitsu Chuo Hospital /ID# 246684, Kisarazu-shi, Chiba
  - Chiba West General Hospital /ID# 230208, Matsudo-shi, Chiba
  - Keyaki Total Clinic /ID# 229648, Matsudo-shi, Chiba
  - Matsudo City Hospital /ID# 232348, Matsudo-shi, Chiba
  - New Tokyo Clinic /ID# 252577, Matsudo-shi, Chiba
  - Hata Orthopaedic Clinic /ID# 258356, Nagareyama-shi, Chiba
  - Japanese Red Cross Narita Hospital /ID# 226738, Narita-shi, Chiba
  - Noda Hospital /ID# 224992, Noda, Chiba
  - Noda Nanbu Clinic /ID# 258353, Noda, Chiba
  - Juntendo University Urayasu Hospital /ID# 226737, Urayasu-shi, Chiba
  - Ishigamiseikei Riumachi Clinic /ID# 238492, Yachiyo, Chiba
  - National Hospital Organization Shimoshizu National Hospital /ID# 250202, Yotsukaido-shi, Chiba
  - Yamada Rheumatology Clinic /ID# 232302, Matsuyama, Ehime
  - Dogo Onsen Hospital /ID# 225755, Matsuyama, Ehime
  - Matsuyama Red Cross Hospital /ID# 226741, Matsuyama, Ehime
  - Jyuzen General Hospital /ID# 249523, Niihama, Ehime
  - Sumitomo Besshi Hospital /ID# 225847, Niihama-shi, Ehime
  - Kuri Orthopedic Clinic /ID# 246724, Shikokuchuo-shi, Ehime
  - Ehime University Hospital /ID# 230277, Toon-shi, Ehime
  - JCHO Uwajima Hospital /ID# 227440, Uwajima-shi, Ehime
  - NHO Awara Hospital /ID# 233863, Awara, Fukui
  - Sugimoto Rheumatology and Internal Medicine Clinic /ID# 224564, Fukui-shi, Fukui
  - Fukuiken Saiseikai Hospital /ID# 243780, Fukui-shi, Fukui
  - Fukui Katsuyama General Hospital /ID# 238739, Katsuyama-shi, Fukui
  - Ota Hospital /ID# 240656, Nyu-gun, Fukui
  - Municipal Tsuruga Hospital /ID# 224472, Tsuruga-shi, Fukui
  - Tochikukai Tochiku Hospital /ID# 239147, Fukuoka, Fukuoka
  - Kondo Clinic for Rheumatism & Orthopedics /ID# 225756, Fukuoka, Fukuoka
  - Hamanomachi Hospital /ID# 239149, Fukuoka, Fukuoka
  - National Hospital Organization Kyushu Medical Center /ID# 239727, Fukuoka, Fukuoka
  - PS Clinic /ID# 223268, Fukuoka, Fukuoka
  - Yagi Hospital - Fukuoka /ID# 223251, Fukuoka, Fukuoka
  - Kyushu University Hospital /ID# 226734, Fukuoka, Fukuoka
  - Kyushu University Hospital /ID# 232147, Fukuoka, Fukuoka
  - Haradoi Hospital /ID# 267424, Fukuoka, Fukuoka
  - Chihaya Hospital /ID# 232522, Fukuoka, Fukuoka
  - Shono Rheumatism Clinic /ID# 232341, Fukuoka, Fukuoka
  - Ogata Orthopedic Clinic /ID# 248098, Fukuoka, Fukuoka
  - Sata Hospital /ID# 225333, Fukuoka, Fukuoka
  - Kyushu Central Hospital of the Mutual Aid Association of Public School Teachers /ID# 233971, Fukuoka, Fukuoka
  - Himeno Hospital /ID# 225340, Hirokawa, Fukuoka
  - Saiseikai Iizuka Kaho Hospital /ID# 246021, Iizuka-shi, Fukuoka
  - Aso Iizuka Hospital /ID# 239148, Iizuka-shi, Fukuoka
  - Aso Iizuka Hospital /ID# 254442, Iizuka-shi, Fukuoka
  - Hiroshima Orthopedic Surgical Clinic /ID# 226830, Kasuya-gun, Fukuoka
  - Kitakyushu Hospital /ID# 262913, Kitakyushu, Fukuoka
  - Kashiwagi Clinic /ID# 246681, Kitakyushu, Fukuoka
  - Yamasu Orthopedic Rheumatic Clinic /ID# 238597, Kitakyushu, Fukuoka
  - Shinkokura Hospital /ID# 225338, Kitakyushu, Fukuoka
  - Hashiguchi Orthopedic Clinic /ID# 245813, Kitakyushu, Fukuoka
  - JR Kyushu Hospital /ID# 225871, Kitakyushu-shi, Fukuoka
  - Kunou Orthopedic Clinic /ID# 226733, Kitakyushu-shi, Fukuoka
  - Kitakyushu Municipal Medical Center /ID# 238574, Kitakyushu-shi, Fukuoka
  - Kenwakai Otemachi Hospital /ID# 250258, Kitakyushu-shi, Fukuoka
  - Kurosaki Orthopedic Hospital /ID# 246026, Kitakyushu-shi, Fukuoka
  - Showa Namiki Hospital /ID# 255156, Kitakyushu-shi, Fukuoka
  - Matsumoto Internal medicine Clinic /ID# 229021, Kitakyushu-shi, Fukuoka
  - Hospital Of The University Of Occupational And Environmental Health, Japan /ID# 224973, Kitakyushu-shi, Fukuoka
  - Wakamatsu Hospital /ID# 230216, Kitakyusyu-shi, Fukuoka
  - Nakamura Orthopedic Surgical Clinic /ID# 232146, Middle City, Fukuoka
  - Obase Hospital /ID# 233846, Miyako-gun, Fukuoka
  - Munakata Medical Association Hospital /ID# 233847, Munakata-shi, Fukuoka
  - Katsuno Orthopaedic and Rehabilitation Department /ID# 224193, Nishiku, Fukuoka
  - Fukuoka Yutaka Central Hospital /ID# 227441, Nogata-shi, Fukuoka
  - Fukuoka Shion Hospital /ID# 232588, Ogōri, Fukuoka
  - Nagata Orthopedic Hospital /ID# 226855, Omuta-shi, Fukuoka
  - Zaitsu Orthopedics Clinic /ID# 258357, Onojo-shi, Fukuoka
  - Nishio Municipal Hospital /ID# 238575, 直方市, Fukuoka
  - Apio Riumachi Clinic /ID# 250257, Aizu-Wakamatsu, Fukushima
  - Fujita General Hospital /ID# 258333, Date-gun, Fukushima
  - Fukushima Medical University Hospital /ID# 231708, Fukushima, Fukushima
  - Yago Rheum Clinic /ID# 227642, Fukushima, Fukushima
  - Jusendo General Hospital /ID# 233885, Koriyama-shi, Fukushima
  - Southern Tohoku Res Inst Neuro /ID# 241923, Koriyama-shi, Fukushima
  - Southern Tohoku Daini Hospital /ID# 240623, Kōriyama, Fukushima
  - Nishimaki Clinic /ID# 238582, Sukagawa, Fukushima
  - Saito Clinic /ID# 238598, 会津若松市, Fukushima
  - Gifu Municipal Hospital /ID# 225837, Gifu, Gifu
  - Ohashi & Tani Orthopedic Clinic /ID# 225863, Gifu, Gifu
  - Kato Internal Medicine Pediatrics /ID# 241161, Gifu, Gifu
  - Gifu Prefectural General Medical Center /ID# 224475, Gifu, Gifu
  - Gifu University Hospital /ID# 230285, Gifu, Gifu
  - Gifu University Hospital /ID# 232499, Gifu, Gifu
  - Gifu University Hospital /ID# 246725, Gifu, Gifu
  - Nagara Orthopedic Clinic /ID# 242030, Gifu, Gifu
  - Gujo City Hospital /ID# 231753, Gujō, Gifu
  - Kaizu Medical Association Hospital /ID# 231725, Kaizu-shi, Gifu
  - Ikeda Clinic /ID# 245097, Kakamigahara, Gifu
  - Kani Tono Hospital /ID# 241154, Kani-shi, Gifu
  - Ota Medical Clinic /ID# 245094, Minokamo, Gifu
  - Ota Hospital /ID# 247770, Minokamo-shi, Gifu
  - Takeda Family Clinic /ID# 267422, Nishikaiden, Gifu
  - Okuda Orthopedic Clinic /ID# 224460, Ogaki-shi, Gifu
  - Kikuike Orthopedic Surgical Clinic /ID# 224988, Seki-shi, Gifu
  - Taguchi Medical Clinic /ID# 260731, Seki-shi, Gifu
  - Duplicate_Chuno Kosei Hospital /ID# 248809, Sekimachi, Gifu
  - Gifu Prefectural Tajimi Hosp /ID# 229656, Tajimi-shi, Gifu
  - Takayama Red Cross Hospital /ID# 252179, Takayama, Gifu
  - Yamamoto Orthopedic Clinic /ID# 233961, Yamagata, Gifu
  - Kusunoki Hospital /ID# 250840, Fujioka, Gunma
  - Takayanagi Seikeigeka Shika Clinic /ID# 238585, Isesaki, Gunma
  - Ishii Hospital /ID# 240618, Isesaki-shi, Gunma
  - Isesaki Fukushima Hospital /ID# 227448, Isesaki-shi, Gunma
  - Jomo Ohashi Clinic /ID# 224993, Maebashi, Gunma
  - Nishida Orthopedics /ID# 223261, Maebashi, Gunma
  - Gunma University Hospital /ID# 243686, Maebashi, Gunma
  - Higashi Maebashi Orthopedic Surgery /ID# 254474, Maebashi, Gunma
  - Takekoshi Clinic /ID# 245814, Ora-gun, Gunma
  - Aozora Orthopedic Rheumatic Clinic /ID# 244226, Ota-shi, Gunma
  - Koiso Clinic /ID# 225335, Ota-shi, Gunma
  - Inoue Hospital /ID# 231714, Takasaki-shi, Gunma
  - Akagi Clinic /ID# 232579, Takasaki-shi, Gunma
  - Keiyu Orthopedic Surgical Clinic /ID# 232581, Tatebayashi-shi, Gunma
  - Okada Orthopedic Clinic /ID# 263046, Tatebayashi-shi, Gunma
  - Mazda Hospital /ID# 239044, Aki-gun, Hiroshima
  - Yoshida General Hospital /ID# 233905, Aki-takata, Hiroshima
  - Numakuma Hospital /ID# 240955, Fukuyama, Hiroshima
  - Ota Memorial Hospital - Fukuyama (Brain Attack Center) /ID# 252211, Fukuyama-shi, Hiroshima
  - JA Hiroshima General Hospital /ID# 244114, Hatsukaichi-shi, Hiroshima
  - Hiroshima Rheumatology Clinic /ID# 230215, Hiroshima, Hiroshima
  - Hiroshima Clinic /ID# 254486, Hiroshima, Hiroshima
  - Hiroshima City Hiroshima Citizens Hospital /ID# 230265, Hiroshima, Hiroshima
  - Hiroshima City Hiroshima Citizens Hospital /ID# 239034, Hiroshima, Hiroshima
  - Hiroshima Red Cross Hospital & Atomic-bomb Survivors Hospital /ID# 238873, Hiroshima, Hiroshima
  - Yamasaki Orthopedic Surgical Clinic /ID# 231748, Hiroshima, Hiroshima
  - Asaminami Clinic /ID# 229644, Hiroshima, Hiroshima
  - Shigenobu Clinic /ID# 232143, Hiroshima, Hiroshima
  - Hiroshima Clinic /ID# 227636, Hiroshima, Hiroshima
  - Hiroshima University Hospital /ID# 232144, Hiroshima, Hiroshima
  - Okita Intenal Medicine Clinic /ID# 232295, Hiroshima, Hiroshima
  - Hashimoto Clinic /ID# 238639, Hiroshima, Hiroshima
  - National Hospital Organization Kure Medical Center /ID# 255154, Kure-shi, Hiroshima
  - Niitani Clinic /ID# 225334, Kure-shi, Hiroshima
  - Kure Kyosai Hospital /ID# 240620, Kure-shi, Hiroshima
  - Kousei General Hospital - Mihara /ID# 275123, Mihara, Hiroshima
  - Hakuryuko Clinics /ID# 244225, Mihara, Hiroshima
  - Mihara Red Cross Hospital /ID# 238594, Mihara-shi, Hiroshima
  - Kousei General Hospital /ID# 224111, Mihara-shi, Hiroshima
  - Miyoshi Central Hospital /ID# 238736, Miyoshi-shi, Hiroshima
  - Seo Clinic /ID# 255161, Sera-gun, Hiroshima
  - Usuki Clinic /ID# 249519, Asahikawa, Hokkaido
  - National Hospital Organization Asahikawa Medical Center /ID# 224415, Asahikawa-shi, Hokkaido
  - Katayama Orthopedic Rheumatology Clinic /ID# 223997, Asahikawa-shi, Hokkaido
  - Asahikawa Medical University Hospital /ID# 232578, Asahikawa-shi, Hokkaido
  - Takeda Orthopedic Clinic /ID# 233909, Ebetsu, Hokkaido
  - Naito Clinic /ID# 238579, Ebetsu, Hokkaido
  - Ebetsu Tanifuji Hospital /ID# 233970, Ebetsu, Hokkaido
  - Furano Hospital /ID# 261290, Furano-shi, Hokkaido
  - Hakodate Red Cross Hospital /ID# 241155, Hakodate, Hokkaido
  - Donan Rheumatism Orthopedic Surgery /ID# 241744, Hakodate, Hokkaido
  - Yunokawa Hot Spring Orthopedic Surgical Clinic /ID# 244228, Hakodate, Hokkaido
  - Yagihara Orthopedic Clinic /ID# 233958, Hakodate Hakodate City, Hokkaido
  - Miyazaki Sei Int Med Clinic /ID# 222604, Hakodate-shi, Hokkaido
  - Hakodate Goryokaku Hospital /ID# 238737, Hakodate-shi, Hokkaido
  - Kitami Red Cross Hospital /ID# 232150, Kitami-shi, Hokkaido
  - Kobayashi Hospital - Kitami /ID# 254484, Kitami-shi, Hokkaido
  - Mombetsu Hospital /ID# 229030, Mombetsu-shi, Hokkaido
  - Tokachi Kinikyo Obihiro Hospital /ID# 248733, Obihiro, Hokkaido
  - Obihiro kosei Hospital /ID# 232344, Obihiro-shi, Hokkaido
  - Omotonaika Clinic /ID# 245807, Otaru, Hokkaido
  - Hokkaido Orthopedics Memorial Hospital /ID# 229646, Sappori-shi, Hokkaido
  - Oshima Internal Medicine and Gastroenterology Clinic /ID# 238470, Sapporo, Hokkaido
  - Sapporo Hokushin Hospital /ID# 241873, Sapporo, Hokkaido
  - Teine Inazumi Hospital /ID# 245073, Sapporo, Hokkaido
  - Kin-ikyo Chuo Hospital /ID# 239039, Sapporo, Hokkaido
  - KKR Sapporo Medical Center Tonan Hospital /ID# 232576, Sapporo, Hokkaido
  - Sagawa Akira Rheumatology Clin /ID# 233860, Sapporo, Hokkaido
  - Soen Central Hospital /ID# 245095, Sapporo, Hokkaido
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital /ID# 241875, Sapporo, Hokkaido
  - JR Sapporo Hospital /ID# 238877, Sapporo, Hokkaido
  - Sapporo Medical Center NTT EC /ID# 238876, Sapporo, Hokkaido
  - Sapporo Rheumatology and immunology clinic /ID# 233861, Sapporo, Hokkaido
  - Sapporo Medical University Hospital /ID# 225851, Sapporo, Hokkaido
  - Sapporo Medical University Hospital /ID# 233857, Sapporo, Hokkaido
  - Sapporo City General Hospital /ID# 240914, Sapporo, Hokkaido
  - Hokkaido University Hospital /ID# 224933, Sapporo, Hokkaido
  - Hokkaido Medical Center /ID# 257002, Sapporo, Hokkaido
  - Hokkaido Medical Center For Rheumatic Diseases /ID# 223274, Sapporo, Hokkaido
  - Sapporo Nishi Maruyama Hospital /ID# 251008, Sapporo, Hokkaido
  - Miyoka internal medicine Clinic /ID# 259338, Sapporo, Hokkaido
  - Clark Hospital /ID# 232590, Sapporo, Hokkaido
  - Takikawa Municipal Hospital /ID# 231713, Takikawa-shi, Hokkaido
  - Yoshikawa Clinic /ID# 233957, Tomakomai, Hokkaido
  - Oki Medical Clinic /ID# 222339, Tomakomai-shi, Hokkaido
  - Wakkanai City Hospital /ID# 243764, Wakkanai, Hokkaido
  - Amagasaki Medical Coop Hospital /ID# 238468, Amagasaki, Hyōgo
  - Kitatsuji Clinic /ID# 225330, Amagasaki-shi, Hyōgo
  - Hyogo Prefectural Amagasaki General Medical Center /ID# 238735, Amagasaki-shi, Hyōgo
  - Matsushima Orthopaedic Clinic /ID# 224106, Amagasaki-shi, Hyōgo
  - Ashiya St. Maria Hospital /ID# 241061, Ashiya, Hyōgo
  - Ando Orthopedic Clinic /ID# 230279, Ashiya, Hyōgo
  - Fujisaki Orthopaedic Clinic /ID# 222337, Ashiya-shi, Hyōgo
  - Jyounan Tago Hospital /ID# 241060, Himeji, Hyōgo
  - Jinno Hospital /ID# 239154, Himeji, Hyōgo
  - Himeji St.Mary's Hospital /ID# 263043, Himeji-shi, Hyōgo
  - Hyogo Prefectural Harima-Himeji General Medical Center /ID# 251720, Himeji-shi, Hyōgo
  - Himeji Medical Center /ID# 225771, Himeji-shi, Hyōgo
  - Himeji Medical Center /ID# 239397, Himeji-shi, Hyōgo
  - Takemura Orthopaedic Clinic /ID# 252181, Himeji-shi, Hyōgo
  - Muroi Medical Office /ID# 243685, Ibo-gun, Hyōgo
  - Ojima Clinic /ID# 239199, Itami, Hyōgo
  - Kinki Central Hospital /ID# 251723, Itami-shi, Hyōgo
  - Itami City Hospital /ID# 240607, Itami-shi, Hyōgo
  - Kakogawa Central City Hospital /ID# 224931, Kakogawa-shi, Hyōgo
  - Konan Kakogawa Hospital /ID# 224196, Kakogawa-shi, Hyōgo
  - Hyogo Prefectural Kakogawa Medical Center /ID# 231722, Kakogawa-shi, Hyōgo
  - Matsubara Mayflower Hospital /ID# 222613, Kato-shi, Hyōgo
  - Harada Rheumatology and Orthopedics Clinic /ID# 225341, Kawanishi-shi, Hyōgo
  - Taketomi Clinic /ID# 261249, Kobe, Hyōgo
  - Kobe University Hospital /ID# 225850, Kobe, Hyōgo
  - Kobe University Hospital /ID# 229028, Kobe, Hyōgo
  - Kobe University Hospital /ID# 231704, Kobe, Hyōgo
  - Kobe City Medical Center General Hospital /ID# 239043, Kobe, Hyōgo
  - Hyogo Prefectural Central Rehabilitation Hospital /ID# 231705, Kobe, Hyōgo
  - Kobe City Medical Center West /ID# 224971, Kobe, Hyōgo
  - Morinobu Clinic /ID# 239729, Kobe, Hyōgo
  - Ichise Clinic /ID# 270444, Kobe, Hyōgo
  - Kobe Kaisei Hospital /ID# 224932, Kobe, Hyōgo
  - Tsuji Rheumatism and Medicine /ID# 229027, Kobe, Hyōgo
  - Konan Medical Center /ID# 224949, Kobe, Hyōgo
  - Matsubara Clinic /ID# 233956, Matsusaka, Hyōgo
  - Nakabayashi Hospital /ID# 233968, Minamiawaji, Hyōgo
  - Yokoyama Orthopaedic Clinic /ID# 223253, Nishinomiya-shi, Hyōgo
  - Nishinomiya Kyoritsu Neurosurgical Hospital /ID# 233955, Nishinomiya-shi, Hyōgo
  - Ohno Clinic /ID# 227445, Nishinomiya-shi, Hyōgo
  - Hyogo Medical University Hospital /ID# 230214, Nishinomiya-shi, Hyōgo
  - Kitano Orthopedic & Surgery Clinic /ID# 238578, Ono-shi, Hyōgo
  - Fukushima Clinic /ID# 256178, Sanda-shi, Hyōgo
  - Takarazuka City Hospital /ID# 239728, Takarazuka-shi, Hyōgo
  - Kodama Hospital /ID# 223252, Takarazuka-shi, Hyōgo
  - Takasago Municipal Hospital /ID# 275666, Takasago, Hyōgo
  - Hyogo Prefectural Tamba Medical Center /ID# 225772, Tamba-shi, Hyōgo
  - Fujiyama Internal Medicine Clinic /ID# 249518, Hitachi-Naka, Ibaraki
  - Hitachinaka General Hospital /ID# 225326, Hitachi-Naka, Ibaraki
  - Oasis Clinic /ID# 225852, Hitachi-shi, Ibaraki
  - Hakujuji General Hospital /ID# 239398, Kamisu, Ibaraki
  - Clinic Quest For Rheumatology & Well Being /ID# 232589, Mito, Ibaraki
  - Moriya Daiichi General Hospital /ID# 241163, Moriya-shi, Ibaraki
  - Namegata District General Hospital /ID# 271891, Namegata, Ibaraki
  - Omitama City Medical Center /ID# 244222, Omitama-shi, Ibaraki
  - Ibaraki Seinan Medical Center Hospital /ID# 246003, Sashima-gun, Ibaraki
  - JA Toride Medical Center /ID# 250201, Toride-shi, Ibaraki
  - Tsuchiura Kyodo General Hospital /ID# 252175, Tsuchiura-shi, Ibaraki
  - Tsukuba Gakuen Hospital /ID# 224197, Tsukuba, Ibaraki
  - University of Tsukuba Hospital /ID# 232346, Tsukuba, Ibaraki
  - Kaga Medical Center /ID# 240627, Kaga, Ishikawa-ken
  - Kanazawa Medical University Hospital /ID# 267425, Kahoku-gun, Ishikawa-ken
  - Saiseikai Kanazawa Hospital /ID# 248736, Kanazawa, Ishikawa-ken
  - Fujita Rheumatic Clinic /ID# 231746, Kanazawa, Ishikawa-ken
  - Ishikawa Prefectural Central Hospital /ID# 244100, Kanazawa, Ishikawa-ken
  - Kanazawa University Hospital /ID# 232500, Kanazawa, Ishikawa-ken
  - Noto General Hospital /ID# 238531, Nanao-shi, Ishikawa-ken
  - Houju Memorial Hospital /ID# 226836, Nomi-shi, Ishikawa-ken
  - Kanazawa Medical University Hospital /ID# 238593, Uchinada-cho, Ishikawa-ken
  - Saito Clinic /ID# 262911, Hanamaki-shi, Iwate
  - Yoshida Orthopaedic Rheumatic /ID# 222609, Morioka, Iwate
  - Komagamine Rheum Ortho Clinic /ID# 223998, Morioka, Iwate
  - Malios Kobayashi Medical Clinic /ID# 265628, Morioka, Iwate
  - Keyaki Clinic /ID# 232504, Morioka, Iwate
  - Shirasawa Orthopeadic Clinic /ID# 259346, Morioka, Iwate
  - Kagawa University Hospital /ID# 225846, Kita-gun, Kagawa-ken
  - Hirose Orthopedic Surgical Clinic /ID# 247876, Marugame, Kagawa-ken
  - Sanuki Municipal Hospital /ID# 224001, Sanuki-shi, Kagawa-ken
  - Otsuka Orthopeadic Clinic /ID# 261287, Takamatsu, Kagawa-ken
  - Sangonoumi Orthopedic Surgical Clinic /ID# 250250, Takamatsu, Kagawa-ken
  - Kagawa Prefectural Central Hospital /ID# 248097, Takamatsu, Kagawa-ken
  - Takamatsu Heiwa Hospital /ID# 240890, Takamatsu, Kagawa-ken
  - Nitta Orthopedic Clinic /ID# 245359, Takamatsu, Kagawa-ken
  - Matsui Hospital /ID# 250254, 観音寺市, Kagawa-ken
  - Yamano Clinic /ID# 233902, Aira, Kagoshima-ken
  - Maehara General Medical Hospital /ID# 256206, Hioki-shi, Kagoshima-ken
  - Higashi Clinic /ID# 253169, Izumi-shi, Kagoshima-ken
  - Uemura Hospital /ID# 275234, Kagoshima, Kagoshima-ken
  - Shiraishi Hospital /ID# 252185, Kagoshima, Kagoshima-ken
  - EIRAKU Internal Medicine Clinic /ID# 233851, Kagoshima, Kagoshima-ken
  - Imamura General Hospital /ID# 232199, Kagoshima, Kagoshima-ken
  - Imamura General Hospital /ID# 234005, Kagoshima, Kagoshima-ken
  - Nakashima Clinic /ID# 252588, Kagoshima, Kagoshima-ken
  - Ueyama Hospital /ID# 231702, Kagoshima, Kagoshima-ken
  - Kagoshima University Hospital /ID# 227442, Kagoshima, Kagoshima-ken
  - Uchimura Orthopedic Clinic /ID# 231749, Kagoshima, Kagoshima-ken
  - Shunyoukai Central Hospital /ID# 259345, Kimotsuki-gun, Kagoshima-ken
  - Nakagawa Seikei Clinic /ID# 222335, Kirishima-shi, Kagoshima-ken
  - Yoshitama Clinic Rheumatology and Internal Medicine /ID# 224195, Kirishima-shi, Kagoshima-ken
  - Wakamatsu Memorial Hospital /ID# 245809, Sendai, Kagoshima-ken
  - Hirata Orthopedic Surgeon Clinic /ID# 245808, 出水市, Kagoshima-ken
  - Oshima Medical Association Hospital /ID# 240628, 奄美市, Kagoshima-ken
  - Kanagawa Prefectural Ashigarakami Hospital /ID# 250207, Ashigarakami, Kanagawa
  - Suzuki Clinic /ID# 232591, Atsugi, Kanagawa
  - Atsugi Nakamachi Clinic /ID# 230260, Atsugi-shi, Kanagawa
  - Mitsuhashi Orthopedics & Rehabilitation Clinic /ID# 229650, Atsugi-shi, Kanagawa
  - Shonan Rhematology Clinic /ID# 233959, Chigasaki-shi, Kanagawa
  - Adachi Masanori Clinic /ID# 225832, Fujisawa-shi, Kanagawa
  - Ikegami Orthopedic Clinic /ID# 226834, Fujisawa-shi, Kanagawa
  - Fujita Clinic /ID# 259348, Fujisawa-shi, Kanagawa
  - Shonan Central Hospital /ID# 251006, Fujisawa-shi, Kanagawa
  - Kinoshita Orthopedic Clinic /ID# 252578, Fujisawa-shi, Kanagawa
  - Fujisawa City Hospital /ID# 227453, Fujisawa-shi, Kanagawa
  - Shonan Daiichi Hospital /ID# 254475, Fujisawa-shi, Kanagawa
  - Takeuchi Orthopedic Clinic /ID# 227629, Fujisawa-shi, Kanagawa
  - Hiratsuka Kyosai Hospital /ID# 230220, Hiratsuka-shi, Kanagawa
  - Tokai University Hospital /ID# 250841, Isehara, Kanagawa
  - Akara Clinic /ID# 250999, Kamakura-shi, Kanagawa
  - Shonan Kamakura General Hospital /ID# 248807, Kamakura-shi, Kanagawa
  - Munehiro Hospital /ID# 229102, Kanazawa-shi, Kanagawa
  - Kawasaki Orthopedic Clinic /ID# 266778, Kawasaki-shi, Kanagawa
  - Kawasaki Municipal Hospital /ID# 222607, Kawasaki-shi, Kanagawa
  - Kawasaki Municipal Ida Hospital /ID# 248770, Kawasaki-shi, Kanagawa
  - Nippon Medical School Musashi Kosugi Hospital /ID# 233880, Kawasaki-shi, Kanagawa
  - Toranomon Hospital Kajigaya /ID# 225833, Kawasaki-shi, Kanagawa
  - Hikarichuo Clinic /ID# 222589, Kawasaki-shi, Kanagawa
  - St Marianna University School Of Medicine /ID# 230261, Kawasaki-shi, Kanagawa
  - Sagami Seikyo Hospital /ID# 244731, Sagamihara, Kanagawa
  - Park Square Clinic /ID# 226839, Sagamihara-shi, Kanagawa
  - Kitasato University Hospital /ID# 224935, Sagamihara-shi, Kanagawa
  - Sagamihara Kyodo Hospital /ID# 231709, Sagamihara-shi, Kanagawa
  - Minamiyamato Hospital /ID# 224451, Yamato-shi, Kanagawa
  - Akizuki Clinic /ID# 225834, Yokohama, Kanagawa
  - Yokohama Municipal Citizen's Hospital /ID# 225874, Yokohama, Kanagawa
  - Ayumi Clinic /ID# 244104, Yokohama, Kanagawa
  - Saiseikai Yokohamashi Tobu /ID# 226828, Yokohama, Kanagawa
  - Yokohama City Minato Red Cross Hospital /ID# 239040, Yokohama, Kanagawa
  - Saiseikai Kanagawaken Hospital /ID# 229653, Yokohama, Kanagawa
  - Ueda Medical Clinic /ID# 231710, Yokohama, Kanagawa
  - Yokohama City University Medical Center /ID# 232351, Yokohama, Kanagawa
  - Yokohama City University Medical Center /ID# 233855, Yokohama, Kanagawa
  - Yokohama Riumachi Clinic /ID# 224938, Yokohama, Kanagawa
  - Saiseikai Yokohamashi Nanbu Hospital /ID# 248808, Yokohama, Kanagawa
  - Sumita Kids Clinic /ID# 238569, Yokohama, Kanagawa
  - Yasoda Orthopedic Rheumatology Clinic /ID# 227628, Yokohama, Kanagawa
  - Yokohama City University Hospital /ID# 232248, Yokohama, Kanagawa
  - Yokohama City University Hospital /ID# 240933, Yokohama, Kanagawa
  - Yokohama City University Hospital /ID# 252599, Yokohama, Kanagawa
  - Yokohama Minami Kyousai Hosp /ID# 227643, Yokohama, Kanagawa
  - Ishizue Orthopedic Clinic /ID# 225865, Yokohama, Kanagawa
  - National Hospital Organization Yokohama Medical Center /ID# 233875, Yokohama, Kanagawa
  - St. Joseph's Hospital /ID# 227452, Yokosuka-shi, Kanagawa
  - Yokosuka Genrl Hospital Uwamachi /ID# 238588, Yokosuka-shi, Kanagawa
  - Kurihamazaitaku Clinic /ID# 257006, Yokosuka-shi, Kanagawa
  - Yokosuka City Hospital /ID# 257003, Yokosuka-shi, Kanagawa
  - Kang Rheuma and Ortho Clinic /ID# 252210, Zushi-shi, Kanagawa
  - Minamiyamatokoza Clinic /ID# 233962, 大和市, Kanagawa
  - WEST Bone Joint clinic /ID# 244103, Agawa-gun, Kochi
  - Machida Clinic /ID# 252593, Agawa-gun, Kochi
  - Usuikai Tano Hospital /ID# 253170, Aki-gun, Kochi
  - East Marine Clinic /ID# 230211, Aki-shi, Kochi
  - Tamaki Clinic /ID# 230263, Kochi, Kochi
  - Bay Side Misato Medical Center /ID# 223266, Kochi, Kochi
  - Kochi Medical School Hospital /ID# 229019, Nankoku-shi, Kochi
  - Nakamura Hospital /ID# 224562, Shimanto-shi, Kochi
  - Genyukai Yoshii Hospital /ID# 226732, Shimanto-shi, Kochi
  - Kikuyochubu Clinic /ID# 251721, Kikuchi-gun, Kumamoto
  - Kumamoto University Hospital /ID# 231718, Kumamoto, Kumamoto
  - Kumamoto University Hospital /ID# 233890, Kumamoto, Kumamoto
  - Kumamoto Orthopaedic Hospital /ID# 232148, Kumamoto, Kumamoto
  - Fujiwara Clinic /ID# 239396, Yamaga, Kumamoto
  - Yamaga Medical Center /ID# 252182, Yamaga-shi, Kumamoto
  - Shiga Clinic /ID# 224109, Ayabe-shi, Kyoto
  - Kyoto Renaiss Hospital /ID# 251719, Fukuchiyama, Kyoto
  - Fukuchiyama City Hospital /ID# 233883, Fukuchiyama-shi, Kyoto
  - Kyoto Okamoto Memorial Hospital /ID# 243741, Kuse-gun, Kyoto
  - Kyoto Okamoto Memorial Hospital /ID# 252597, Kuse-gun, Kyoto
  - Takeda Hospital /ID# 224954, Kyoto, Kyoto
  - JyuJyo Takeda Rehabilitation /ID# 233858, Kyoto, Kyoto
  - Japanese Red Cross Kyoto Daini Hospital /ID# 241922, Kyoto, Kyoto
  - Kamigyo Clinic /ID# 225844, Kyoto, Kyoto
  - University Hospital Kyoto Prefectural University of Medicine /ID# 239038, Kyoto, Kyoto
  - Japanese Red Cross Kyoto Daiichi Hosital /ID# 239192, Kyoto, Kyoto
  - Japanese Red Cross Kyoto Daiichi Hosital /ID# 239350, Kyoto, Kyoto
  - Rakuyo Hospital /ID# 241062, Kyoto, Kyoto
  - Kyoto University Hospital /ID# 224930, Kyoto, Kyoto
  - Kyoto University Hospital /ID# 238874, Kyoto, Kyoto
  - Rakuwakai Otowa Hosptial /ID# 230266, Kyoto, Kyoto
  - National Hospital Organization Kyoto Medical Center /ID# 225853, Kyoto, Kyoto
  - National Hospital Organization Utano National Hospital /ID# 223994, Kyoto, Kyoto
  - Komuro Orthopaedic Clinic /ID# 229162, Kyoto, Kyoto
  - Kyoto Tanabe Central Hospital /ID# 239392, Kyōtanabe, Kyoto
  - Fujii Obaku Station Clinic /ID# 242022, Uji, Kyoto
  - Kawamoto Orthopedic Surgical Clinic /ID# 240621, Uji, Kyoto
  - Matsui Orthopedics Clinic /ID# 232149, Uji-shi, Kyoto
  - Uji Takeda Hospital /ID# 251007, Uji-shi, Kyoto
  - Uji Tokushukai Medical Center /ID# 244211, Uji-shi, Kyoto
  - Nakajima Clinic /ID# 240617, Yawata, Kyoto
  - Morita Orthopedic Surgical Clinic /ID# 243719, Ise, Mie-ken
  - Ise Rheumatology Hand Clinic /ID# 229163, Ise-shi, Mie-ken
  - Kuwana city medical center /ID# 225875, Kuwana-shi, Mie-ken
  - Otsuji Orthopedic Clinic /ID# 226835, Matsusaka-shi, Mie-ken
  - National Mie Hospital /ID# 241871, Tsu, Mie-ken
  - Uemura Orthopaedic Surgery /ID# 238601, Tsu, Mie-ken
  - Higuchi Orthopedic Clinic /ID# 239393, Tsu, Mie-ken
  - Matsumotokaido Clinic /ID# 241874, Yokkaichi, Mie-ken
  - Yokkaichi Hazu Medical Center /ID# 224014, Yokkaichi-shi, Mie-ken
  - Tomidahama Hospital /ID# 239348, Yokkaichi-shi, Mie-ken
  - Tomidahama Hospital /ID# 275667, Yokkaichi-shi, Mie-ken
  - Mori Orthopedic Surgery Clinic /ID# 250995, Iwanuma, Miyagi
  - Ishibashi Hospital - Kurihara /ID# 240609, Kurihara-shi, Miyagi
  - Kurokawa Hospital /ID# 243776, Kurokawa-gun, Miyagi
  - Osaki Citizen Hospital /ID# 231706, Osaki-shi, Miyagi
  - Ogura Orthopaedic Surgery /ID# 232501, Sendai, Miyagi
  - IMS Meirikai Sendai General Hospital /ID# 232193, Sendai, Miyagi
  - Tohoku University Hospital /ID# 232345, Sendai, Miyagi
  - Tohoku University Hospital /ID# 239150, Sendai, Miyagi
  - Blue Sky Clinic /ID# 240619, Sendai, Miyagi
  - Honma Memorial Tohoku Orthopedic Surgery / Tohoku Dental /ID# 241266, Sendai, Miyagi
  - Izumi Himawari Clinic /ID# 225776, Sendai, Miyagi
  - Tohoku Rosai Hospital /ID# 238538, Sendai, Miyagi
  - Tohoku Medical and Pharmaceuti /ID# 233865, Sendai, Miyagi
  - Hikarigaoka Spellman Hospital /ID# 226736, Sendai, Miyagi
  - Munakata Yasuhiko Clinic /ID# 233948, Sendai, Miyagi
  - Shishido Clinic /ID# 238734, 東松島市, Miyagi
  - Matsuyama Clinic /ID# 241157, Capital City, Miyazaki
  - Keimei Memorial Hospital /ID# 225869, Higashimorokata, Miyazaki
  - Miyazaki Saiseikai Hyuga Hospital /ID# 250256, Higashiusuki-gun, Miyazaki
  - Chiyoda Hospital /ID# 226758, Hyuga-shi, Miyazaki
  - Ikei Hospital /ID# 248099, Kobayashi, Miyazaki
  - Kusumoto Clinic /ID# 251714, Kobayashi-shi, Miyazaki
  - Nojiri Central Hospital /ID# 246027, Kobayashi-shi, Miyazaki
  - Ikenoue Orthopedic Clinic /ID# 251004, Miyakonojo-shi, Miyazaki
  - Miyakonojo National Hospital /ID# 233850, Miyakonojo-shi, Miyazaki
  - Miyanaga Hospital /ID# 240657, Miyakonojō, Miyazaki
  - Medical Corporation Keiai Kai Clinic /ID# 232342, Miyazaki, Miyazaki
  - Shishime Orthopedics Hospital /ID# 250199, Miyazaki, Miyazaki
  - Zenjinkai Shimin-no-mori Hospital /ID# 225303, Miyazaki, Miyazaki
  - University of Miyazaki Hospital /ID# 225766, Miyazaki, Miyazaki
  - University of Miyazaki Hospital /ID# 252173, Miyazaki, Miyazaki
  - Siloam Internal Medicine Clinic /ID# 255160, Nichinan-shi, Miyazaki
  - Nobeoka Medical Association Hospital /ID# 244221, Nobeoka, Miyazaki
  - Yanazawa Orthopedic Clinic /ID# 233954, Nobeoka-shi, Miyazaki
  - Sanzai Hospital /ID# 238596, West City, Miyazaki
  - Iida Hospital /ID# 279004, Iida, Nagano
  - Marunouchi Hospital /ID# 231711, Matsumoto-shi, Nagano
  - Shinshu University Hospital /ID# 232200, Matsumoto-shi, Nagano
  - Shinonoi General Hospital /ID# 233887, Nagano, Nagano
  - Saku Central Hospital /ID# 239031, Saku-shi, Nagano
  - Asama General Hospital /ID# 238603, Saku-shi, Nagano
  - Nagasaki Goto Chuoh Hospital /ID# 229160, Goto-shi, Nagasaki
  - Suga Orthopedic Hospital /ID# 241153, Isahaya-shi, Nagasaki
  - Duplicate_Isahaya Health Insurance General Hospital /ID# 233849, Isahaya-shi, Nagasaki
  - Nagasaki Medical Hospital Rheumatology /ID# 224563, Nagasaki, Nagasaki
  - Takahara Chuou Clinic /ID# 262028, Nagasaki, Nagasaki
  - Wajinkai Hospital /ID# 229108, Nagasaki, Nagasaki
  - Tsukazaki Clinic /ID# 231752, Nagasaki, Nagasaki
  - Jap Red Cross Nagasaki Genbaku /ID# 233848, Nagasaki, Nagasaki
  - Aino Memorial Hospital /ID# 233908, Nagasaki, Nagasaki
  - Miyashita Rheumatology Clinic /ID# 241159, Omura-shi, Nagasaki
  - Sasebo Chuo Hospital /ID# 224002, Sasebo-shi, Nagasaki
  - Inada Orthopedic Surgical Clinic /ID# 242021, Shimabara, Nagasaki
  - Matsuoka Hospital /ID# 225302, Shimabara-shi, Nagasaki
  - Nagasaki Kita Hospital /ID# 229024, Togitsu, Nagasaki
  - Ikoma City Hospital /ID# 258345, Ikoma-shi, Nara
  - Nara Hospital Kinki University Faculty of Medicine, /ID# 233891, Ikoma-shi, Nara
  - Kanshiba Asahigaoka Hospital /ID# 232570, Kanshiba-shi, Nara
  - Nijoekimae Clinic /ID# 227447, Kashiba-shi, Nara
  - Higami Hospital /ID# 224012, Kashihara-shi, Nara
  - Nara Medical University Hospital /ID# 224414, Kashihara-shi, Nara
  - Nara Medical University Hospital /ID# 243773, Kashihara-shi, Nara
  - Nampei Clinic /ID# 230281, Katsuragi-shi, Nara
  - Hara Orthopaedic Clinic /ID# 245093, Kitakōriyamachō, Nara
  - Nara City Hospital /ID# 249527, Nara, Nara
  - Nishinokyo Hospital /ID# 250247, Nara, Nara
  - Sawai Hospital /ID# 238599, Nara, Nara
  - Harada Clinic /ID# 240651, Nara, Nara
  - Tomio Clinic /ID# 231747, Nara, Nara
  - Kokuho Chuo Hospital /ID# 244102, Tawaramoto, Nara
  - Tenri Hospital /ID# 224929, Tenri-shi, Nara
  - Ninomiya Orthopedic Clinic /ID# 238532, Yamatotakada-shi, Nara
  - Minami Nara General Medical Center /ID# 244096, Yoshino-gun, Nara
  - Katsumi Seikei /ID# 223306, Chuo-ku, Niigata
  - Niigata Prefectural Ctr Hosp /ID# 227625, Jōetsu, Niigata
  - Ii Internal Medicine Clinic /ID# 246004, Jōetsu, Niigata
  - Minamiuonuma City Hospital /ID# 252575, Minamiuonuma-shi, Niigata
  - Yukiguni Yamato City Hospital /ID# 232515, Minamiuonuma-shi, Niigata
  - Mitsuke City Hospital /ID# 232502, Mitsuke, Niigata
  - Aile Home Clinic /ID# 244109, Nagaoka, Niigata
  - Nagaoka Chuo General Hospital /ID# 268875, Nagaoka, Niigata
  - Aile Home Clinic Nagaoka /ID# 266780, Nagaoka-shi, Niigata
  - Nagaoka Red Cross Hospital /ID# 229046, Nagaoka-shi, Niigata
  - Kimura Orthopedic Clinic /ID# 248773, Niigata, Niigata
  - Saiseikai Niigata Hospital /ID# 232585, Niigata, Niigata
  - Niigata Medical Center /ID# 262026, Niigata, Niigata
  - NHO Nishiniigata Chuo Hospital /ID# 267371, Niigata, Niigata
  - Niigata University Medical & Dental Hospital /ID# 239030, Niigata, Niigata
  - Niigata University Medical & Dental Hospital /ID# 239033, Niigata, Niigata
  - Doya Rehabilitation & Orthopedic Clinic /ID# 268348, Niigata, Niigata
  - Sakai Family Clinic /ID# 251695, Tsubame-shi, Niigata
  - National Hospital Organization Beppu Medical Center /ID# 225339, Beppu-shi, Oita Prefecture
  - Kyushu University Beppu Hospital /ID# 224413, Beppu-shi, Oita Prefecture
  - Kawashima Orthopaedic Hospital /ID# 241918, Nakatsu, Oita Prefecture
  - Sakai Hospital /ID# 229114, Nakatsu-shi, Oita Prefecture
  - Oita Red Cross Hospital /ID# 223250, Ōita, Oita Prefecture
  - Akeno Central Hospital /ID# 225870, Ōita, Oita Prefecture
  - Oita Medical Center /ID# 246002, Ōita, Oita Prefecture
  - Sato Daiichi Hospital /ID# 242031, Usa-shi, Oita Prefecture
  - Usuki Cosmos Hospital /ID# 252590, Usuki-shi, Oita Prefecture
  - Kurashiki Central Hospital Riverside /ID# 248782, Kurashiki, Okayama-ken
  - Kurashiki Sweet Hospital /ID# 223249, Kurashiki-shi, Okayama-ken
  - Kurashiki Heisei Hospital /ID# 230075, Kurashiki-shi, Okayama-ken
  - Kurashiki Central Hospital /ID# 231701, Kurashiki-shi, Okayama-ken
  - Kurashiki Municipal Hospital /ID# 242395, Kurashiki-shi, Okayama-ken
  - Mizushima Kyodo Hospital /ID# 239035, Kurashiki-shi, Okayama-ken
  - Okayama Saiseikai Outpatient Center Hospital /ID# 241742, Okayama, Okayama-ken
  - Okayama Central Hospital /ID# 262688, Okayama, Okayama-ken
  - Okayama University Hospital /ID# 225337, Okayama, Okayama-ken
  - Okayama University Hospital /ID# 226740, Okayama, Okayama-ken
  - Tsuyama Daiichi Hospital /ID# 233895, Tsuyama, Okayama-ken
  - Shinkenko Clinic /ID# 246657, Naha, Okinawa
  - Oura Clinic /ID# 223273, Naha, Okinawa
  - Naha City Hospital /ID# 248806, Naha, Okinawa
  - Shurijo Jokamachi Clinic Daiichi /ID# 238576, Naha, Okinawa
  - Miyara Clinic /ID# 251694, Naha, Okinawa
  - Chibana Clinic /ID# 250994, Okinawa-shi, Okinawa
  - Yaesekai Dojin Hospital /ID# 226829, Urasoe-shi, Okinawa
  - Araya Clinic /ID# 253171, Daito-shi, Osaka
  - Osaka Minami Coop Clinic /ID# 231751, Habikino, Osaka
  - Masuda Orthopedic Surgical Clinic /ID# 262687, Habikino-shi, Osaka
  - Choshi Clinic /ID# 250843, Habikino-shi, Osaka
  - Osaka Habikino Medical Center /ID# 244110, Habikino-shi, Osaka
  - Tanaka Clinic /ID# 244730, Hannan-shi, Osaka
  - Mori Clinic /ID# 244206, Higashiosaka, Osaka
  - Sobajima Clinic /ID# 252584, Higashiosaka-shi, Osaka
  - Shigematsu Orthopaedic & Hand Clinic /ID# 252576, Higashiosaka-shi, Osaka
  - Yamaguchi Clinic /ID# 225327, Higashiosaka-shi, Osaka
  - Kosugi Orthopedic Rheumatology /ID# 230262, Higashiosaka-shi, Osaka
  - Kaneko Orthopaedic Clinic /ID# 229109, Higashiosaka-shi, Osaka
  - Shiomi Orthopedic Clinic /ID# 223255, Higashiosaka-shi, Osaka
  - Higashiosaka City Medical Center /ID# 232571, Higashiosaka-shi, Osaka
  - Hirakata Kohsai Hospital /ID# 243058, Hirakata, Osaka
  - Negi Orthopedic Surgeon and Rheumatology Clinic /ID# 244101, Hirakata, Osaka
  - Nagisa Umeda Orthopaedic Clinic /ID# 238537, Hirakata, Osaka
  - Hoshigaoka Medical Center /ID# 225864, Hirakata-shi, Osaka
  - Kansai Medical University Hospital /ID# 232523, Hirakata-shi, Osaka
  - Arisawa General Hospital /ID# 224936, Hirakata-shi, Osaka
  - North Osaka Housenka Hospital /ID# 245092, Ibaraki, Osaka
  - Kunisato Orthopedic Surgical Clinic /ID# 244115, Ibaraki-shi, Osaka
  - Yamaguchi Clinic /ID# 252574, Ibaraki-shi, Osaka
  - Santa Maria Hospital /ID# 224476, Ibaraki-shi, Osaka
  - Sugimoto Clinic /ID# 225872, Ikeda-shi, Osaka
  - Izumi City General Hospital /ID# 225768, Izumi-shi, Osaka
  - Arita Orthopedic Surgical Clinic /ID# 224481, Izumisano, Osaka
  - Rinku General Medical Center /ID# 227639, Izumisano, Osaka
  - Rinku General Medical Center /ID# 273570, Izumisano, Osaka
  - Kayashimaikuno Hospital /ID# 273568, Kadoma, Osaka
  - Maki Rehabilitation Hospital /ID# 272715, Kadoma-shi, Osaka
  - Kaizuka City Hospital /ID# 243684, Kaizuka-shi, Osaka
  - Kashiwara Municipal Hospital /ID# 244108, Kashihara, Osaka
  - Kanemoto Orthopaedics Clinic /ID# 226816, Kashiwara-shi, Osaka
  - Kitada Clinic /ID# 252212, Katano-shi, Osaka
  - National Hospital Organization Osaka Minami Medical Center /ID# 225770, Kawachinagano Shi, Osaka
  - Kusumoto Clinic /ID# 248101, Kawachinagano-shi, Osaka
  - Kishiwada Tokushukai Hospital /ID# 244204, Kishiwada-shi, Osaka
  - Kishiwada City Hospital /ID# 232587, Kishiwada-shi, Osaka
  - Kishiwada City Hospital /ID# 240653, Kishiwada-shi, Osaka
  - Kishiwada City Hospital /ID# 243742, Kishiwada-shi, Osaka
  - Inoue Orthopedics & Qastrointestinal Clinic /ID# 251002, Matsubara, Osaka
  - Ikeshita Orthopedic Surgical Clinic /ID# 267426, Matsubara-shi, Osaka
  - Mino City Hospital /ID# 229161, Minoh, Osaka
  - Hakuto Clinic /ID# 231754, Minoh, Osaka
  - Ishii Seikeigeka Clinic /ID# 224986, Minoo-shi, Osaka
  - Moriguchi Ikuno Memorial Hospital /ID# 267421, Moriguchi-shi, Osaka
  - Kawamoto Clinic /ID# 271697, Moriguchi-shi, Osaka
  - Osaka Hospital /ID# 223258, Neyagawa, Osaka
  - Sumitomo Hospital /ID# 230207, Osaka, Osaka
  - Kinshukai Infusion Clinic /ID# 225757, Osaka, Osaka
  - Osaka Saiseikai Nakatsu Hospital /ID# 229026, Osaka, Osaka
  - Kitano Hospital, Tazuke Kofukai Medical Research Institute /ID# 227638, Osaka, Osaka
  - Ushio Clinic /ID# 224006, Osaka, Osaka
  - Touei Clinic /ID# 224482, Osaka, Osaka
  - Yodogawa Christian Hospital /ID# 225867, Osaka, Osaka
  - Osaka City General Hospital /ID# 225306, Osaka, Osaka
  - Osaka City General Hospital /ID# 240912, Osaka, Osaka
  - Osaka City General Hospital /ID# 258326, Osaka, Osaka
  - Saijo Clinic /ID# 231729, Osaka, Osaka
  - Omori Orthopedic Surgical Clinic /ID# 273569, Osaka, Osaka
  - Coop Osaka Hospital /ID# 275119, Osaka, Osaka
  - Hinata Clinic /ID# 264436, Osaka, Osaka
  - Hayaishi Hospital /ID# 225305, Osaka, Osaka
  - Uehonmachi Riumachi Komachi Clinic /ID# 241063, Osaka, Osaka
  - Okada Clinic /ID# 270951, Osaka, Osaka
  - Osaka Red Cross Hospital /ID# 232343, Osaka, Osaka
  - Daini Osaka Police Hospital /ID# 229025, Osaka, Osaka
  - Shirasaki Orthopedic Clinic /ID# 240652, Osaka, Osaka
  - Yoshida Orthopedic Clinic /ID# 240658, Osaka, Osaka
  - Kanayama Internal Medicine Clinic /ID# 240654, Osaka, Osaka
  - Shinto Orthopaedic Rheumatic Clinic /ID# 231721, Osaka, Osaka
  - Osaka General Hospital of Japan West Railway Company /ID# 242398, Osaka, Osaka
  - Osaka Metropolitan University Hospital /ID# 224003, Osaka, Osaka
  - Osaka Metropolitan University Hospital /ID# 240608, Osaka, Osaka
  - Koryokai Hospital /ID# 251709, Osaka, Osaka
  - Kansai Denryoku Hospital /ID# 240616, Osaka, Osaka
  - Nakanoshima Iwaki Orthopedic Clinic /ID# 263044, Osaka, Osaka
  - Osaka Social Medical Center Hospital /ID# 244105, Osaka, Osaka
  - Daiwa Chuo Hospital /ID# 258349, Osaka, Osaka
  - Yamamoto Third Hospital /ID# 231727, Osaka, Osaka
  - Osaka General Medical Center /ID# 223270, Osaka, Osaka
  - Minamiosaka Hospital /ID# 254485, Osaka, Osaka
  - Minamiosaka Hospital /ID# 258342, Osaka, Osaka
  - Sakurakai Hospital /ID# 229660, Osakasayama-shi, Osaka
  - Kashimoto Hospital /ID# 252594, Osakasayama-shi, Osaka
  - Seigakai Tsujimoto Hospital /ID# 267427, Osakasayama-shi, Osaka
  - Kindai University Hospital /ID# 225343, Osakasayama-shi, Osaka
  - Asakayama General Hospital /ID# 250255, Sakai, Osaka
  - Osada Orthopedic Surgeon Clinic /ID# 233966, Sakai, Osaka
  - Hino Clinic - Sakai /ID# 275630, Sakai, Osaka
  - Duplicate_Sakai Sakibana Hospital /ID# 225873, Sakai-shi, Osaka
  - Hankai Hospital /ID# 225767, Sakai-shi, Osaka
  - Osaka Rosai Hospital /ID# 241122, Sakai-shi, Osaka
  - Mitani Family Clinic /ID# 252596, Sakai-shi, Osaka
  - Nagayama Rheumatology Orthopaedics /ID# 222478, Sakai-shi, Osaka
  - Sakai Heisei Hospital /ID# 252213, Sakai-shi, Osaka
  - Bellland General Hospital /ID# 261289, Sakai-shi, Osaka
  - Nogami Senshu Rehabilitation Clinic /ID# 267423, Sennan-shi, Osaka
  - Kyowakai Hospital /ID# 226759, Suita-shi, Osaka
  - Yoshida Clinic /ID# 224989, Suita-shi, Osaka
  - Osaka Saiseikai Senri Hospital /ID# 229645, Suita-shi, Osaka
  - The University of Osaka Hospital /ID# 227444, Suita-shi, Osaka
  - The University of Osaka Hospital /ID# 238577, Suita-shi, Osaka
  - The University of Osaka Hospital /ID# 242028, Suita-shi, Osaka
  - Saito Seikeigeka /ID# 222612, Taisho-ku, Osaka
  - Nagainaika Clinic /ID# 238539, Takatsuki, Osaka
  - Osaka Medical and Pharmaceutical University Hospital /ID# 231743, Takatsuki-shi, Osaka
  - Osaka Saiseikai Tondabayashi Hospital /ID# 262910, Tondabayashi-shi, Osaka
  - Toyonaka Keijinkai Hospital /ID# 231742, Toyonaka, Osaka
  - Kataoka Orthopedics & Reumatology /ID# 233898, Toyonaka, Osaka
  - Asai Orthopedic Clinic /ID# 225332, Toyonaka-shi, Osaka
  - Ando Orthopaedic Clinic /ID# 225308, Toyonaka-shi, Osaka
  - Toyonaka Municipal Hospital /ID# 249398, Toyonaka-shi, Osaka
  - Kansai Medical Hospital /ID# 241817, Toyonaka-shi, Osaka
  - National Hospital Organization Osaka Toneyama Medical Center /ID# 227443, Toyonaka-shi, Osaka
  - Nakatani Orthopedic Surgical Clinic /ID# 238600, Yao, Osaka
  - Ishinkai Yao Rehabilitation Hospital /ID# 252592, Yao-shi, Osaka
  - Ojima Orthopedic Clinic /ID# 240624, 高石市, Osaka
  - You-You Clinic /ID# 240626, Karatsu, Saga-ken
  - Kawaguchi Orthopedic Surgical Clinic /ID# 230286, Karatsu-shi, Saga-ken
  - Kamiarita Orthopedic Clinic /ID# 226827, Nishimatsuura-gun, Saga-ken
  - Hiramatsu Hospital /ID# 241152, Ogi-shi, Saga-ken
  - Tanaka Hospital /ID# 223308, Saga, Saga-ken
  - Magokoro Clinic /ID# 246682, Tosu, Saga-ken
  - Suzuki Clinic /ID# 260343, Asaka-shi, Saitama
  - Fukaya Red Cross Hospital /ID# 231723, Fukaya-shi, Saitama
  - Higashimatsuyama Medical Association Hospital /ID# 251711, Higashimatsuyama-shi, Saitama
  - Kono Orthop. and Int. Medical Clinic /ID# 224423, Higashimatsuyama-shi, Saitama
  - Ohno Clinic /ID# 230287, Hiki-gun, Saitama
  - Saitama Medical University Hospital /ID# 226739, Iruma-gun, Saitama
  - IMS Miyoshi General Hospital /ID# 242167, Iruma-gun, Saitama
  - Toyooka Daiichi Hospital /ID# 231717, Iruma-shi, Saitama
  - Shuuwa General Hospital /ID# 233964, Kasukabe, Saitama
  - Ogawa Internal Medicine Clinic - Kawagoe /ID# 238493, Kawagoe, Saitama
  - Saitama Medical Center /ID# 225868, Kawagoe, Saitama
  - Sekishindo Hospital /ID# 231715, Kawagoe-shi, Saitama
  - Sekishindo Hospital /ID# 233872, Kawagoe-shi, Saitama
  - Nagasawa Clinic /ID# 232349, Kawagoe-shi, Saitama
  - Ishii Orthopedics Clinic /ID# 229159, Kawaguchi-shi, Saitama
  - Saiseikai Kawaguchi General Hospital /ID# 238570, Kawaguchi-shi, Saitama
  - Kaneko Clinic - Kawaguchi /ID# 222343, Kawaguchi-shi, Saitama
  - Nakada Hospital /ID# 224601, Kazo-shi, Saitama
  - Matsuzaki Orthopaedics and Rheumatology Clinic /ID# 229041, Kitamoto, Saitama
  - Kitasato University Medical Center /ID# 239045, Kitamoto-shi, Saitama
  - Shinkuki General Hospital /ID# 254487, Kuki-shi, Saitama
  - Kuki Medical Clinic /ID# 261288, Kuki-shi, Saitama
  - Kumagaya General Hospital /ID# 233856, Kumagaya-shi, Saitama
  - Toma Hospital /ID# 224937, Kumagaya-shi, Saitama
  - Niiza Shiki Central General Hospital /ID# 241839, Niiza, Saitama
  - Suda Orthopaedic Clinic /ID# 225336, Niiza-shi, Saitama
  - Duplicate_Aoki Medical Clinic /ID# 225830, Saitama-shi, Saitama
  - Japanese Red Cross Saitama Hospital /ID# 232195, Saitama-shi, Saitama
  - Wakaba Hospital /ID# 241816, Sakado-shi, Saitama
  - Azuma Rheumatology Clinic /ID# 222587, Sayama-shi, Saitama
  - Tanaka Orthopedic Clinic /ID# 231728, Shiki-shi, Saitama
  - Sato Saitama Rheumatoid Clinic /ID# 245091, Toda, Saitama
  - Tokorozawa Central Hospital /ID# 243688, Tokorozawa, Saitama
  - Hirose Clinic - Tokorozawa /ID# 224972, Tokorozawa-shi, Saitama
  - Duplicate_Hara Kids Clinic /ID# 252579, Tokorozawa-shi, Saitama
  - Kanetsu Hospital /ID# 240915, Tsurugashima-shi, Saitama
  - Mami Clinic of Internal Medicine /ID# 240932, ふじみ野市, Saitama
  - Karimoto Seikeigeka Clinic /ID# 224101, Gamou-gun, Shiga
  - Hikone Chuo Hospital /ID# 244230, Hikone, Shiga
  - Municipal Nagahama Hospital /ID# 238469, Nagahama, Shiga
  - Oumi Rheumatology Clinic /ID# 248737, Ōmihachiman, Shiga
  - Yura Clinic /ID# 249515, Ōtsu, Shiga
  - Sakamoto Democratic Clinic /ID# 232260, Ōtsu, Shiga
  - Japanese Red Cross Otsu Shiga Hospital /ID# 233859, Ōtsu, Shiga
  - Japanese Red Cross Otsu Shiga Hospital /ID# 252184, Ōtsu, Shiga
  - Shiga University of Medical Science Hospital /ID# 242396, Ōtsu, Shiga
  - Ōtsu Red Cross Hospital /ID# 243761, Ōtsu, Shiga
  - Nakamura Clinic /ID# 225845, Hamada-shi, Shimane
  - Sugiura Clinic /ID# 224192, Izumo-shi, Shimane
  - Shimane University Hospital /ID# 238573, Izumo-shi, Shimane
  - Matsue Red Cross Hospital /ID# 254483, Matsue, Shimane
  - Oda Municipal Hospital /ID# 244094, Oda, Shimane
  - Unnan City Hospital /ID# 265626, Unnan-shi, Shimane
  - Kawanishi Clinic /ID# 227626, Atami-shi, Shizuoka
  - Fujieda Municipal General Hospital /ID# 232196, Fujieda-shi, Shizuoka
  - Naito Orthopedic Surgical Clinic /ID# 224987, Fujinomiya-shi, Shizuoka
  - Kobayakawa Orthopedic & Rheumatologic Clinic /ID# 252177, Fukuroi-shi, Shizuoka
  - Fukuma Clinic /ID# 239400, Hamamatsu, Shizuoka
  - Hamamatsu South Hospital /ID# 222584, Hamamatsu, Shizuoka
  - Hayakawa Clinic - Hammatsu /ID# 231724, Hamamatsu, Shizuoka
  - Ja Shizuoka Kohseiren Enshu Hospital /ID# 266779, Hamamatsu, Shizuoka
  - Hamamatsu University Hospital /ID# 238590, Hamamatsu, Shizuoka
  - Hamamatsu University Hospital /ID# 244729, Hamamatsu, Shizuoka
  - Yasuhiro Clinic /ID# 225329, Hamamatsu, Shizuoka
  - Suzukake Central Hospital /ID# 257005, Hamamatsu, Shizuoka
  - Hamamatsu Medical Center /ID# 239349, Hamamatsu, Shizuoka
  - Fujiwara Orthopedic Clinic /ID# 240615, Hamamatsu, Shizuoka
  - Kobori Orthopedic Clinic /ID# 225346, Hamamatsu, Shizuoka
  - Kimoto Clinic /ID# 248734, Hamamatsu, Shizuoka
  - Hokuto Wakaba Hospital /ID# 256194, Hamamatsu, Shizuoka
  - Nisizaka Orthopedic Clinic /ID# 222590, Hamamatsu, Shizuoka
  - Futaba Clinic /ID# 241158, Iwata-shi, Shizuoka
  - Juntendo University Shizuoka Hospital /ID# 224453, Izunokuni-shi, Shizuoka
  - Koide Clinic /ID# 247878, Kosai, Shizuoka
  - Ohara Internal Medicine Rheumatic Clinic /ID# 243689, Shizuoka, Shizuoka
  - Japanese Red Cross Shizuoka Hospital /ID# 224939, Shizuoka, Shizuoka
  - Miyake Clinic of Orthopedic Surgery /ID# 223307, Shizuoka, Shizuoka
  - Shizuoka Saiseikai Genaral Hospital /ID# 225835, Shizuoka, Shizuoka
  - Matsuuraseikei /ID# 225836, Shizuoka, Shizuoka
  - Kusanagi Seikei Clinic /ID# 224452, Shizuoka, Shizuoka
  - Koga Community Hospital /ID# 251681, Yaizu, Shizuoka
  - Imai Hospital /ID# 232194, Ashikaga, Tochigi
  - Satsuki Home Clinic Mashiko /ID# 240953, Haga-gun, Tochigi
  - Dokkyo Medical University Hospital /ID# 233852, Mibu, Tochigi
  - Kawamura Internal Medicine Clinic /ID# 225839, Oyama-shi, Tochigi
  - Kokubunji Sakura Clinic /ID# 227449, Shimotsuke, Tochigi
  - Jichi Medical University Hospital /ID# 229034, Shimotsuke-shi, Tochigi
  - Tochigi Medical Center Shimotsuga /ID# 238584, Tochigi-shi, Tochigi
  - Takase Orthopedic Clinic /ID# 241872, Utsunomiya, Tochigi
  - Yukawanaika Clinic /ID# 224199, Utsunomiya, Tochigi
  - Deiriumachikanaika Clinic /ID# 239151, Utsunomiya, Tochigi
  - Tochigi Rheumatology Clinic /ID# 238583, Utsunomiya, Tochigi
  - Utsunomiya Central Clinic /ID# 233969, Utsunomiya, Tochigi
  - National Hospital Organization Utsunomiya Hospital /ID# 227641, Utsunomiya, Tochigi
  - Anan Medical Center /ID# 224103, Anan-shi, Tokushima
  - Tokushima Prefectural Kaifu Hospital /ID# 238742, Kaifugun, Tokushima
  - Kunimi Clinic /ID# 225331, Mima-shi, Tokushima
  - Kondo Hospital /ID# 238571, Tokushima, Tokushima
  - Seihou-kai Mima Hospital /ID# 232145, Yoshinogawa-shi, Tokushima
  - Yamaji Clinic /ID# 232582, Adachi City, Tokyo
  - Adachikeiyu Orthopedic Surgical Clinic /ID# 233963, Adachi Ward, Tokyo
  - Tokyo Kousei Hospital /ID# 224102, Adachi-ku, Tokyo
  - Haijima Yamakami Clinic /ID# 248768, Akishima, Tokyo
  - Akishima Hospital /ID# 239347, Akishima, Tokyo
  - Akishima Rhematology Clinic /ID# 233950, Akishima, Tokyo
  - Nishiogu RA Clinic /ID# 238733, Arakawa-ku, Tokyo
  - Juntendo University Hospital /ID# 225328, Bunkyo-ku, Tokyo
  - Institute of Science Tokyo Hospital /ID# 224934, Bunkyo-ku, Tokyo
  - Nippon Medical School Hospital /ID# 229649, Bunkyo-ku, Tokyo
  - The University of Tokyo Hospital /ID# 224424, Bunkyo-ku, Tokyo
  - The University of Tokyo Hospital /ID# 251697, Bunkyo-ku, Tokyo
  - Yamanaka Clinic /ID# 256188, Chiyoda-ku, Tokyo
  - Mitsui Memorial Hospital /ID# 230218, Chiyoda-ku, Tokyo
  - Chofu Touzan Hospital /ID# 227631, Chofu-shi, Tokyo
  - Suzuki Clinic Orthopaedics River City /ID# 259340, Chuo-ku, Tokyo
  - St. Lukes International Hospital /ID# 224419, Chuo-ku, Tokyo
  - Tsukiji Immuno-Rheumatology Clinic /ID# 248810, Chuo-shi, Tokyo
  - Keyakinamiki?Orthopedics /ID# 233901, Fuchū, Tokyo
  - Ando Surgical Internal Medicine Clinic /ID# 231750, Hachiōji, Tokyo
  - Tama-Hokubu Medical Center /ID# 225876, Higashimurayama-shi, Tokyo
  - Tokyo Metropolitan Geriatric /ID# 252595, Itabashi-ku, Tokyo
  - Negishi Orthopedic Clinic /ID# 231757, Itabashi-ku, Tokyo
  - Koto Hospital /ID# 260208, Jiangdong District, Tokyo
  - JCHO Tokyo Joto Hospital /ID# 242399, Jiangdong, Tokyo
  - Nankatsu Kanamachi Ophthalmology /ID# 252180, Katsushika-ku, Tokyo
  - Ashizawa Orthopedic Rheumatism Clinic /ID# 251712, Katsushika-ku, Tokyo
  - Otake Clinic /ID# 242020, Kita Ward, Tokyo
  - Takinogawa Hospital /ID# 224473, Kita-ku, Tokyo
  - Shono Orthopedic Clinic /ID# 225344, Kita-ku, Tokyo
  - Fukujuji Hospital /ID# 251724, Kiyose-shi, Tokyo
  - National Hospital Organization Tokyo National Hospital /ID# 233877, Kiyose-shi, Tokyo
  - Kawashima Orthopedic Clinic /ID# 238495, Kodaira, Tokyo
  - Showa University Koto Toyosu Hospital /ID# 226742, Koto-ku, Tokyo
  - Juntendo Tokyo Koto Geriatric Medical Center /ID# 226813, Koto-ku, Tokyo
  - Juntendo Tokyo Koto Geriatric Medical Center /ID# 227630, Koto-ku, Tokyo
  - Ishikawa Medical Clinic /ID# 247877, Machida, Tokyo
  - Machida Municipal Hospital /ID# 238879, Machida-shi, Tokyo
  - Meguro Kakinokizaka Clinic /ID# 232584, Meguro City, Tokyo
  - National Hospital Organization Tokyo Medical Center /ID# 222588, Meguro-ku, Tokyo
  - Toho University Ohashi Medical Center - Tokyo /ID# 233904, Meguro-ku, Tokyo
  - Tokyo Kyosai Hospital /ID# 240942, Meguro-ku, Tokyo
  - Toranomon Hospital /ID# 233886, Minato-ku, Tokyo
  - Kanenaka Neurosurgery Clinic /ID# 252214, Nakano-ku, Tokyo
  - Oedo Orthopedic Surgery and Internal Medicine /ID# 223305, Nerima City, Tokyo
  - Matsuda Orthopedic Rheuma Clinic /ID# 238587, Nerima-ku, Tokyo
  - Juntendo Univ Nerima Hospital /ID# 244099, Nerima-ku, Tokyo
  - Kamiyama Clinic /ID# 226815, Nerima-ku, Tokyo
  - Mitamura Clinic /ID# 250248, Nerima-ku, Tokyo
  - Nerima Hikarigaoka Hospital /ID# 245098, Nerima-ku, Tokyo
  - Kasugacho Clinic /ID# 251005, Nerima-ku, Tokyo
  - Tanaka Clinic /ID# 238589, Nishi-Tokyo-shi, Tokyo
  - Takagi Hospital /ID# 232249, Ōme, Tokyo
  - Ai Medical Clinic /ID# 231744, Ōta-ku, Tokyo
  - Omori Sanno Hospital /ID# 248772, Ōta-ku, Tokyo
  - Toho University Medical Center Omori Hospital /ID# 240625, Ōta-ku, Tokyo
  - Yasuda Seikei Clinic /ID# 222484, Ōta-ku, Tokyo
  - Okazaki Clinic /ID# 239153, Ōta-ku, Tokyo
  - Tokyo Arthritis Clinic /ID# 248100, Ōta-ku, Tokyo
  - Otomo Clinic /ID# 242165, Setagaya City, Tokyo
  - Matsuta Clinic /ID# 229042, Setagaya-ku, Tokyo
  - Setagaya Rheumatic Clinic /ID# 224425, Setagaya-ku, Tokyo
  - Setagaya Rheum Soshigaya Clinic /ID# 260160, Setagaya-ku, Tokyo
  - Soshigaya Okura Clinic /ID# 232583, Setagaya-ku, Tokyo
  - Shinjuku South Rheumatic Clinic /ID# 231719, Shibuya-ku, Tokyo
  - Shinjuku Tsurukame Clinic /ID# 257004, Shibuya-ku, Tokyo
  - Ueda Medical Clinic /ID# 239191, Shinagawa Ward, Tokyo
  - NTT Medical Center Tokyo /ID# 233879, Shinagawa-ku, Tokyo
  - Ebara Home Care Clinic /ID# 258360, Shinagawa-ku, Tokyo
  - Showa University East Hospital /ID# 229892, Shinagawa, Tokyo
  - Hosaka Clinic /ID# 231756, Shinagawa, Tokyo
  - Keio University Hospital /ID# 224013, Shinjuku-ku, Tokyo
  - Tokyo Women's Medical University Hospital /ID# 229045, Shinjuku-ku, Tokyo
  - Tokyo Women's Medical University Hospital /ID# 233874, Shinjuku-ku, Tokyo
  - Japan Community Health care Organization Tokyo Yamate Medical Center /ID# 251725, Shinjuku-ku, Tokyo
  - Nishimura Orthopedic Clinic /ID# 225838, Shinjuku-ku, Tokyo
  - Meiyo Immunology & Rheumatology Clinic /ID# 252186, Suginami -ku, Tokyo
  - Hattori Seikei Clinic /ID# 227632, Suginami-ku, Tokyo
  - Koenji Orthopedic Clinic /ID# 233949, Suginami, Tokyo
  - Ogikubo Clinic /ID# 240650, Suginami, Tokyo
  - Tokyo Skytree Station Medical Clinic /ID# 238872, Sumida Ward, Tokyo
  - Medical Corporation Uchida Clinic /ID# 224418, Sumida-ku, Tokyo
  - Tokyo Metropolitan Bokutoh Hospital /ID# 232350, Sumida-ku, Tokyo
  - Nokubo Orthopedic Clinic /ID# 225841, Tachikawa-shi, Tokyo
  - Inoue Orthopedics Surgery /ID# 243720, Taito-Ku, Tokyo
  - Tokyo Metropolitan Ohtsuka Hos /ID# 242029, Toshima-ku, Tokyo
  - Obayashi Clinic /ID# 243749, Xiaoping, Tokyo
  - Aoyoko Orthopedic Clinic /ID# 240655, 品川区, Tokyo
  - Minami Otsuka Clinic /ID# 241267, 豊島区, Tokyo
  - Takita Orthopedic Clinic /ID# 225765, Yonagi-shi, Tottori
  - Tottori University Hospital /ID# 240606, Yonago-shi, Tottori
  - Tottori University Hospital /ID# 244095, Yonago-shi, Tottori
  - Imizu Municipal Hospital /ID# 238743, Imizu-shi, Toyama
  - Kurobe City Hospital /ID# 239395, Kurobe-shi, Toyama
  - 500koku Orthopedic Clinic /ID# 229103, Nakaniikawa-gun, Toyama
  - Yoshimi Hospital /ID# 233953, Namerikawa-shi, Toyama
  - Takaokaekinan Clinic /ID# 238572, Takaoka, Toyama
  - Takaoka Rheumatic Orthopedic Clinic /ID# 223265, Takaoka-shi, Toyama
  - Tonami General Hospital /ID# 224940, Tonami-shi, Toyama
  - Toyama University Hospital /ID# 224603, Toyama, Toyama
  - Toyama Prefectural Central Hospital /ID# 225307, Toyama, Toyama
  - Sainou Hospital /ID# 229107, Yokoyama-shi, Toyama
  - Kitade Hospital /ID# 239753, Gobo-shi, Wakayama
  - Chuki Clinic /ID# 259342, Gobo-shi, Wakayama
  - Naga municipal Hospital /ID# 240913, Kinokawa, Wakayama
  - Shirahama Hamayu Hospital /ID# 223254, Nishimuro-gun, Wakayama
  - Tsuji Clinic /ID# 229657, Tanabe-shi, Wakayama
  - Social Insurance Kinan Hosp /ID# 252183, Tanabe-shi, Wakayama
  - Saiseikai Wakayama Hospital /ID# 262027, Wakayama, Wakayama
  - Japanese Red Cross Wakayama Medical Center /ID# 233967, Wakayama, Wakayama
  - Kotonoura Rehabilitation Center Hospital /ID# 270115, Wakayama, Wakayama
  - Wakayama Medical University Hospital /ID# 225769, Wakayama, Wakayama
  - Wakayama Medical University Hospital /ID# 243723, Wakayama, Wakayama
  - Jinmachi Clinic /ID# 229735, Higashine-shi, Yamagata
  - Nihonkai General Hospital /ID# 233854, Sakata-shi, Yamagata
  - Yamagata University Hospital /ID# 230284, Yamagata, Yamagata
  - Yamaguchi Grand Medical Center /ID# 229891, Hohu-shi, Yamaguchi
  - Shunan Memorial Hospital /ID# 233842, Kudamatsu-shi, Yamaguchi
  - Nagato General Hospital /ID# 224991, Nagato-shi, Yamaguchi
  - Sanyo-Onoda Municipal Hospital /ID# 266720, Sanyōonoda, Yamaguchi
  - Yamaguchi Rosai Hospital /ID# 248771, Sanyōonoda, Yamaguchi
  - Shimonoseki City Hospital /ID# 226731, Shimonoseki, Yamaguchi
  - Nibu Clinic /ID# 238740, Shimonoseki, Yamaguchi
  - Kawata Junko Clinic /ID# 222611, Shimonoseki-shi, Yamaguchi
  - Tokito Clinic Rheumatology and Orthopaedics Surgery /ID# 224000, Shimonoseki-shi, Yamaguchi
  - Fukuta Clinic /ID# 223248, Ube-shi, Yamaguchi
  - Yamaguchi University Hospital /ID# 225764, Ube-shi, Yamaguchi
  - Yamaguchi University Hospital /ID# 246656, Ube-shi, Yamaguchi
  - Tanekubo Clinic /ID# 241268, Yamaguchi, Yamaguchi
  - Ono clinic For Orthopaedics And Rheumatology /ID# 240938, Yamaguchi, Yamaguchi
  - Yamaguchi Red Cross Hospital /ID# 225311, Yamaguchi, Yamaguchi
  - Shuto General Hospital /ID# 250197, Yanai-shi, Yamaguchi
  - University of Yamanashi Hospital /ID# 233876, Chuo-shi, Yamanashi
  - University of Yamanashi Hospital /ID# 243721, Chuo-shi, Yamanashi
  - Kasugai Clinic /ID# 229661, Fuefuki-shi, Yamanashi
  - Nishioka Clinic RA /ID# 248769, Kofu, Yamanashi
  - Kamiya Orthopedic Clinic /ID# 225345, Kofu, Yamanashi
  - Tsurutoranomongeka Rehabilitation Clinic /ID# 238540, Tsuru, Yamanashi
  - Fukui General Clinic /ID# 239152, Fukui
  - Fukuoka Sports Clinic /ID# 238541, Fukuoka
  - Souseikai Fukuoka Mirai Hospital /ID# 233965, Fukuoka
  - Fukushima Red Cross Hospital /ID# 224417, Fukushima
  - JR Hiroshima Hospital /ID# 265624, Hiroshima
  - Hiroshima Prefecture Hospital /ID# 243683, Hiroshima
  - Izumihara Rheumatic and Medical Clinic /ID# 225849, Kagoshima
  - Sunsun Clinic /ID# 230076, Kochi
  - Kataoka Orthopaedic Surgeon and Rheumatology /ID# 238604, Kumamoto
  - Takeda General Hospital /ID# 238741, Kyoto
  - Yu Family Clinic /ID# 223259, Miyagi
  - Takeuchi Hospital /ID# 245096, Miyazaki
  - Miyazaki Zenjinkai Hospital /ID# 231755, Miyazaki
  - Ikeda Clinic /ID# 242025, Nagano
  - Hayashi Rheumatology Orthopedic Clinic /ID# 224602, Nagano
  - Nagasaki University Hospital /ID# 227637, Nagasaki
  - Jurakukai Ohno Memorial Hospital /ID# 225342, Naniwa
  - Niigata Bandai Hospital /ID# 268873, Niigata
  - Niigata Rinko Hospital /ID# 240613, Niigata
  - Okayama City General Medical Center Okayama City Hospital /ID# 247762, Okayama
  - Higashisumiyoshi Morimoto Hospital /ID# 239726, Osaka
  - Daido Clinic - Osaka /ID# 227446, Osaka
  - Nippon Life Saiseikai Public Interest Foundation Nippon Life Hospital /ID# 251001, Osaka
  - Maeshima Rheumatology Clinic /ID# 224010, Ōita
  - Ome Municipal General Hospital /ID# 264445, Ōme
  - Suzuhiro Clinic /ID# 226837, Saitama
  - Saitama City Hospital /ID# 238738, Saitama
  - Tmg Asaka Medical Center /ID# 230264, Saitama
  - Ina Hospital /ID# 273567, Saitama
  - Takeishi Naika Clinic /ID# 238471, Sano-shi
  - Shimoda Medical Center /ID# 250249, Shimoda
  - Shizuoka Rheumatism Orthopedic Rehabilitation Hospital /ID# 222608, Shizuoka
  - Shizuoka Magarikane Clinic /ID# 238529, Shizuoka
  - Tanaka Hiroya Clinic /ID# 224477, Takarazu-shi
  - IMSUT Hospital, The Institute of Medical Science, The University of Tokyo /ID# 240649, Tokyo
  - Tokyo Women'S Medical University Medical Center East /ID# 238586, Tokyo
  - Tokyo Women'S Medical University Medical Center East /ID# 241265, Tokyo
  - Nissan Tamagawa Hospital /ID# 227450, Tokyo
  - Teikyo University Hospital /ID# 227451, Tokyo
  - Itabashi Central General Hospital /ID# 249528, Tokyo
  - Tottori Prefectural Central Hospital /ID# 278104, Tottori
  - Japanese Red Cross Tottori Hospital /ID# 233845, Tottori
  - Toyama Hospital /ID# 224974, Toyama
  - Yokohama Ekisaikai Hospital /ID# 244218, Yokohama
  - Hyogo Prefectural Awaji Medical Center /ID# 244219, 洲本市

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.rxabbvie.com/